CLINICAL TRIAL: NCT07398248
Title: The Effects of Powerlifting-Based Training on Hormonal, Metabolic, and Lipid Profile Parameters in Athletes: A Randomized Controlled Trial
Brief Title: Effects of Powerlifting-Based Training in Athletes
Acronym: PLBT-ATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ramazan Erdoğan (Other)
Responsible Party: Sponsor-Investigator, Ramazan Erdoğan, Associate Professor, Munzur University
Organization: Munzur University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-31679287-663.05-523405; E-31679287-663.05-523405 (Other: Ethics Committee of Dicle University)
Record Dates: First submitted 2025-12-29; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Physical Fitness; Hormonal Response; Metabolic Parameters
Keywords: Powerlifting; Strength Training; Basketball
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Powerlifting-Based Training Group (Experimental): Participants performed a structured powerlifting-based training program in addition to their regular basketball training. The intervention was conducted three days per week for six weeks. Each session lasted approximately 60 minutes and included a standardized warm-up, a powerlifting-focused main training phase, and a cool-down period.
  The training program emphasized the squat, bench press, and deadlift exercises performed with progressive intensity. Accessory exercises targeting lower-body strength, upper-body musculature, and core stability were included. High-intensity bodyweight exercises were also performed to enhance anaerobic capacity and neuromuscular performance. All training sessions were supervised by qualified staff.
  Interventions: Other: Powerlifting-Based Training; Other: Blood Sampling and Laboratory Analysis
- Control Group (Other): Participants continued their usual basketball training routines throughout the study period without any additional strength or powerlifting-based exercises.
  Interventions: Other: Usual Basketball Training; Other: Blood Sampling and Laboratory Analysis

INTERVENTIONS:
Other: Powerlifting-Based Training — Participants will perform a structured powerlifting-based training program including squat, bench press, and deadlift exercises, conducted 3 sessions per week for 8 weeks under supervision.
  Arms: Powerlifting-Based Training Group
Other: Usual Basketball Training — Participants continued their usual basketball training routines without any additional strength or powerlifting-based exercises.
  Arms: Control Group
Other: Blood Sampling and Laboratory Analysis — Venous blood samples were collected from participants at baseline and post-intervention following an overnight fast. Hormonal parameters were analyzed using ELISA methods, and metabolic and lipid profile parameters were analyzed using an automated biochemical analyzer.

SUMMARY:
This randomized controlled trial aims to examine the effects of a weightlifting-based training program on hormonal, metabolic, and lipid profile parameters in athletes. Participants will be randomly assigned to either a weightlifting-based training group or a control group. The training program will be implemented for a specific period, and relevant blood parameters will be evaluated before and after the intervention. The findings of this study may contribute to a better understanding of the physiological effects of weightlifting-based training on athletes.

DETAILED DESCRIPTION:
This study is designed as a randomized controlled trial to investigate the effects of a structured weightlifting training program on hormonal, metabolic, and lipid profile parameters in athletes. Eligible participants will be randomly assigned to either an intervention group undergoing a weightlifting-based training protocol or a control group continuing their usual training routines.

The intervention will be implemented over a predetermined training period, and outcome measures will include selected hormonal, metabolic, and lipid profile markers obtained from blood samples. Measurements will be taken at baseline and at the end of the training period. The results of this study are expected to provide evidence on physiological adaptations associated with weightlifting-based training and offer practical implications for training program design in athletic populations.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players aged 18 to 24 years
* At least two years of regular sports experience
* Actively participating in basketball training and competition
* Voluntary participation with written informed consent

Exclusion Criteria:

* History of musculoskeletal injury or surgery within the last six months
* Presence of chronic disease or metabolic disorder
* Use of performance-enhancing drugs or hormonal supplements
* Participation in another structured training program during the study period

Ages: 18 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male athletes were eligible to participate in this study.
Enrollment: 30 (Actual)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Mean Change in Fasting Serum Total Testosterone Concentration Measured by ELISA (ng/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum total testosterone concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Serum Cortisol Concentration Measured by ELISA (µg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum cortisol concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Serum Growth Hormone Concentration Measured by ELISA (ng/mL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum growth hormone concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Serum Thyroid-Stimulating Hormone Concentration Measured by ELISA (µIU/mL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum thyroid-stimulating hormone concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Serum Triiodothyronine Concentration Measured by ELISA (ng/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum triiodothyronine concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Serum Thyroxine Concentration Measured by ELISA (µg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum thyroxine concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
Mean Change in Fasting Serum Insulin Concentration Measured by ELISA (µIU/mL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting serum insulin concentrations, measured from venous blood samples using a commercially available enzyme-linked immunosorbent assay (ELISA).
Mean Change in Fasting Blood Glucose Concentration Measured by Automated Biochemical Analyzer (mg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention fasting blood glucose concentrations, measured from venous blood samples using an automated biochemical analyzer.
Mean Change in Total Cholesterol Concentration Measured by Automated Biochemical Analyzer (mg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention total cholesterol concentrations, measured from venous blood samples using an automated biochemical analyzer.
Mean Change in Low-Density Lipoprotein Cholesterol Concentration Measured by Automated Biochemical Analyzer (mg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention low-density lipoprotein cholesterol concentrations, measured from venous blood samples using an automated biochemical analyzer.
Mean Change in High-Density Lipoprotein Cholesterol Concentration Measured by Automated Biochemical Analyzer (mg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention high-density lipoprotein cholesterol concentrations, measured from venous blood samples using an automated biochemical analyzer.
Mean Change in Triglyceride Concentration Measured by Automated Biochemical Analyzer (mg/dL) | Baseline and post-intervention (8 weeks)
  Mean difference between baseline and post-intervention triglyceride concentrations, measured from venous blood samples using an automated biochemical analyzer.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Faculty of Sport Sciences, Tunceli, Center
  - Munzur University, Bitlis, Tunceli

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical restrictions, participant confidentiality concerns, and the absence of participant consent for data sharing beyond the scope of this study.

DOCUMENTS (1):
  • Study Protocol (2025-09-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT07398248/Prot_000.pdf